CLINICAL TRIAL: NCT03967145
Title: Reliability and Validity of the Turkish Version of the Glaucoma Quality of Life-15 Questionnaire
Brief Title: Turkish Version of the Glaucoma Quality of Life-15 Questionnaire
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Collaborators: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Özgül Öztürk, Principal Investigator, Acibadem University
Other Study IDs: ATADEK 2019-7/2
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Glaucoma; Quality of Life
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Determining quality of life — Quality of Life

SUMMARY:
Glaucoma is a disease with irreversible loss of visual field and optic neuropathy and is the most important cause of irreversible vision loss after cataract in the world. Although clinical evaluations reveal the level of glaucoma quantitatively, it is necessary to evaluate the impact of this pathology on daily functions and quality of life with a holistic perspective and to provide appropriate advice to patients according to the information obtained. Glaucoma Quality of Life -15 Questionnaire (GQoL-15) was developed by Nelson et al. in 2003 to evaluate the quality of life of glaucoma patients. The aim of this study is to translate GQoL-15 into Turkish and evaluate its test-retest reliability for Turkish-speaking population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary open angle glaucoma more than 6 months with visual field tests,
* Have the sufficient cognitive level to answer the scale questions.

Exclusion Criteria:

* To have retinal or optic nerve pathologies that may cause loss of visual field or decrease in visual field except glaucoma,
* To undergo eye surgery in the last 3 months.

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Primary Open-Angle Glaucoma patients
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Glaucoma Quality of Life 15 Questionnaire total score | 6 months
  GQoL-15 total score was got after calculate the all subscale values. Subscales are as; 1) Central and near vision (two questions); 2) Peripheral vision (six questions); 3) Dark adaptation (six questions); 4) Outdoor mobility (one question). The item responses for each factor are marked on a five-point scale (1 meaning no difficulty and 5 meaning severe difficulty), 0 is marked if the participant does not perform the activity because of non-visual causes. Higher GQL-15 total scores and subscale scores are reveals lower QoL.
25-item National Eye Institute Visual Functioning Questionnaire (NEI-VFQ 25) | 6 months
  NEI-VFQ 25 total score was got after calculate the all values. It is comprised of 25 items which are; general health and vision, ocular pain, difficulty with vision activities, distance-vision activities, limitation of social functioning, mental health problems, role limitations, dependency on others, driving difficulties, difficulty with color vision and difficulty with peripheral vision. A total score of NEI-VFQ 25 is generated by averaging the scores of all subscales except general health. The item responses for factors are marked on a five or six point scale. Subscale score can be calculated, overall total lower score indicates better vision-related QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Özgül Öztürk, Principal Investigator — Acibadem University
Locations (1):
- Yücel Öztürk, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No